CLINICAL TRIAL: NCT03436433
Title: Phase II Trial of Seizure Prophylaxis in Brain Tumor Patients Undergoing Neurosurgical Procedure
Brief Title: Seizure Prophylaxis in Patients With Glioma or Brain Metastasis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Did not enroll as planned
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00081334
Record Dates: First submitted 2018-02-12; First posted 2018-02-19 (Actual); Results first posted 2021-12-30 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Glioma; Glioma of Brain; Brain Tumor
Keywords: anti-epileptic drugs; seizure prophylaxis; levetiracetam
MeSH Terms: conditions — Glioma; Brain Neoplasms | interventions — Lacosamide; Levetiracetam

STUDY DESIGN:
Intervention Model Description: Upon consent, patients will be randomized in REDCap™ to receive either LCM, LEV, or no AED. Randomization will be stratified by suspected histologic grade (LGG vs HGG vs brain metastasis) based on MRI review by the treating neurosurgeon and/or neuro-oncologist. A stratified permuted block randomization algorithm will be used assign patients to treatment arms.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Lacosamide (Active Comparator): Enrolled subjects will be randomized to receive Lacosamide.
  Interventions: Drug: Lacosamide
- Levetiracetam (Active Comparator): Enrolled subjects will be randomized to receive Levetiracetam.
  Interventions: Drug: Levetiracetam
- No anti-epileptic (No Intervention): Enrolled subjects will be randomized to not receive anti-epileptic drugs.

INTERVENTIONS:
Drug: Lacosamide — LCM 100mg twice a day.
  Other Names: LCM; Vimpat
  Arms: Lacosamide
Drug: Levetiracetam — LEV 1000mg twice a day.
  Other Names: LEV; Keppra
  Arms: Levetiracetam

SUMMARY:
This protocol is designed to assess the need for seizure prophylaxis in the perioperative period for patients undergoing neurosurgical procedure (gross-total resection, sub-total resection or biopsy) for suspected diagnosis of new, recurrent or transformed glioma (WHO grade I-IV) and brain metastasis. This will be determined by observing the impact of Lacosamide (LCM), Levetiracetam (LEV), or no anti-epileptic drug (AED) on whether visits to the emergency department (ED) or hospital re-admissions occur within 30 days after procedure. A secondary endpoint will evaluate the safety and tolerability of LCM and LEV. Exploratory endpoints will evaluate admission duration for the procedure, number of post-operative provider communications (telephone, email, and additional clinic encounters, etc.), and patient risk factors associated with post-operative seizure.

DETAILED DESCRIPTION:
The protocol will assess the need for AED prophylaxis during the post-operative period in patients undergoing neurosurgical procedure for a suspected diagnosis of glioma (WHO grade I-IV) and brain metastasis. Patients (n=116) will be consented and randomized at their pre-operative assessment, either at their pre-operative clinic visit or in the ED, if that is the time of their initial presentation prior to surgery. There will be three arms to the study - patients will be randomized to LCM, LEV, or control (no AED). Randomization will be stratified by suspected grade (LGG vs HGG) and brain metastasis. The AED can be initiated anytime within 48 hours before neurosurgical procedure.

Doses will be either LCM 100mg twice a day (BID) (Arm A), LEV 1000mg BID (Arm B), or no AED (Arm C). If a patient is randomized to Arm C and undergoes tumor mapping, the patient is allowed to receive one dose of AED in the operating room. If a patient is randomized to Arm A or Arm B and takes the morning dose of their AED, they do not need an intra-operative dose of AED. If a patient has a seizure during the post-operative period, AEDs will be adjusted at the discretion of the treating physician. However, if a patient has intolerable side effects, patients will be changed to a different dose of the same medicine before consideration of another AED [i.e., BID to four times a day (QID) dosing if patient experiences diplopia on LCM].

Patients with high-grade tumors (newly-diagnosed or transformed) will be treated with standard radiation and temozolomide therapy per the Stupp protocol 25,70. For these patients, an AED taper will be initiated at the first clinic visit after completion of radiation. For patients with a low-grade tumor or recurrent disease of any grade or brain metastasis, an AED taper will be initiated at the first scheduled post-operative visit, approximately 6-10 weeks after the operation. LCM will be tapered by 100mg a week one week at a time. LEV will be tapered 500-1000mg one week at a time.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a suspected diagnosis of new, recurrent, or transformed glioma (WHO grade I-IV) or brain metastasis scheduled for neurosurgical procedure (gross-total resection, sub-total resection or biopsy) at Duke University Medical Center (DUMC);
2. Safe for surgery per treating neurosurgeon;
3. Due to the potential implications of the treatment on the developing central nervous system (CNS), all patients must be ≥ 18 years of age at the time of entry into the study;
4. Laboratory Studies:

   1. Total bilirubin, Serum Glutamic Oxaloacetic Transaminase (SGOT), Serum Glutamic Pyruvic Transaminase (SGPT), Alkaline Phosphatase (ALK) ≤ 1.5 x upper limit of normal (ULN)
   2. Creatinine ≤ 1.5
5. A signed informed consent form approved by the Duke University Institutional Review Board (IRB) will be required for patient enrollment into the study. Patients must be able to read and understand the informed consent document and must sign the informed consent indicating that they are aware of the investigational nature of this study.
6. Patients of child bearing potential or with partners of child-bearing potential must agree to practice recommended contraceptive methods to prevent pregnancy during treatment and for 1 month after the last dose of AED for women and men.

Exclusion Criteria:

1. Pregnant or need to breast feed during the study period (Negative urine β-human chorionic gonadotropin (HCG) test required), or unable to maintain use of contraception while on study and for 1 month after the last dose of AED;
2. Patients already on AED(s);
3. Known history of epilepsy/seizure disorder;
4. Known history of dependency/abuse of psychopharmaceuticals, alcohol, illicit drugs or narcotics;
5. Any significant medical or psychiatric illness that cannot be adequately controlled with appropriate therapy or would compromise the patient's ability to tolerate therapy, per the discretion of the treating investigator;
6. Known allergy to LCM or LEV.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2019-01-31 (Actual); Primary Completion 2020-12-04 (Actual); Study Completion 2020-12-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Annick Desjardins, M.D., Principal Investigator — Duke University
Locations (1):
- Duke Comprehensive Cancer Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened to accrual on January 31st, 2019. Potential participants were approached and invited to participate in the study during their standard of care medical visits at the Duke Cancer Center (outpatient clinic). Enrollment was suspended during the COVID-19 pandemic, from March to August 2020. The study was finally closed to accrual on February 10, 2021.
Period: Overall Study
Arm/Group | Lacosamide | Levetiracetam | No Anti-epileptic
Started | 1 | 2 | 1
Completed | 1 | 2 | 1
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lacosamide | Levetiracetam | No Anti-epileptic | Total
Number analyzed (Participants) | 1 | 2 | 1 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 41 | 51 (17) | 54 | 49.3 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1 | 2
  Male | 1 | 1 | 0 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Black/African-American | 1 | 0 | 0 | 1
  Race: White/Caucasian | 0 | 2 | 1 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1 | 2 | 1 | 4
Anxiety [Count of Participants; unit: Participants] | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With an ED Visit/Hospital Readmission Within 30 Days of Craniotomy
Description: The primary objective of this study is to assess the impact of LCM, LEV or, no AED in patients undergoing craniotomy for suspected new, recurrent or transformed glioma (WHO Gr I-IV) or brain metastasis on ED visits and readmissions within 30 days of craniotomy.
Time Frame: 30 days following surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Lacosamide | Levetiracetam | No Anti-epileptic
Number analyzed (Participants) | 1 | 2 | 1
Participants | 0 | 0 | 1

2. Secondary Outcome: Number of Participants With an Adverse Event Within First 30 Days After Craniotomy
Description: Adverse events related to LCM, LEV, and no drug within first 30 days after craniotomy.
Time Frame: 30 days following surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Lacosamide | Levetiracetam | No Anti-epileptic
Number analyzed (Participants) | 1 | 2 | 1
Participants
  Dizziness | 1 | 1 | 1
  Somnolence | 1 | 2 | 1
  Cognitive disturbance | 1 | 0 | 1
  Nausea | 1 | 1 | 0
  Vomiting | 1 | 0 | 0
  Ataxia | 1 | 0 | 0
  Suicide thought | 0 | 0 | 0
  Suicide attempt | 0 | 0 | 0
  Anxiety | 1 | 1 | 0
  Depression | 0 | 0 | 0
  Irritability | 1 | 1 | 0
  Psychosis | 0 | 0 | 0
  Personality change | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Lacosamide | Levetiracetam | No Anti-epileptic
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/2 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/2 | 0/1
Other Adverse Events (participants affected / at risk) | 1/1 | 2/2 | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lacosamide (N=1) | Levetiracetam (N=2) | No Anti-epileptic (N=1)
Dizziness (Nervous system disorders) | 1 | 1 | 1
Somnolence (Nervous system disorders) | 1 | 2 | 1
Cognitive disturbance (Nervous system disorders) | 1 | 0 | 1
Nausea (General disorders) | 1 | 1 | 0
Vomiting (General disorders) | 1 | 0 | 0
Ataxia (Nervous system disorders) | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 1 | 0
Irritability (Psychiatric disorders) | 1 | 1 | 0

LIMITATIONS AND CAVEATS:
This study was limited by the small sample size, and a dataset with a larger sample size should be used to further evaluate the impact of LCM, LEV, and no antiepileptic drugs on adverse events, ED visits and hospital readmissions in the future.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2020-08-04): https://cdn.clinicaltrials.gov/large-docs/33/NCT03436433/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-27): https://cdn.clinicaltrials.gov/large-docs/33/NCT03436433/SAP_002.pdf